CLINICAL TRIAL: NCT02526160
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study With Open-Label Extension to Assess the Efficacy and Safety of KRN23 in Adults With X-linked Hypophosphatemia (XLH)
Brief Title: Study of KRN23 in Adults With X-linked Hypophosphatemia (XLH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UX023-CL303; 2014-005529-11 (EudraCT Number)
Expanded Access: NCT03775187 (Available)
Record Dates: First submitted 2015-07-17; First posted 2015-08-18 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: X-linked Hypophosphatemia
Keywords: KRN23; Fibroblast growth factor 23 (FGF23); XLH; X-linked hypophosphatemia; burosumab; Crysvita
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Burosumab 1 mg/kg (Experimental): Burosumab 1 mg/kg administered subcutaneously (SC) every 4 weeks, for the duration of the study.
  Interventions: Biological: burosumab
- Placebo (Placebo Comparator): Placebo administered SC every 4 weeks through Week 24, followed by burosumab 1 mg/kg, for the duration of the study.
  Interventions: Biological: burosumab; Other: Placebo

INTERVENTIONS:
Biological: burosumab — solution for SC injection
  Other Names: UX023; KRN23; Crysvita
Other: Placebo — saline solution for SC injection
  Arms: Placebo

SUMMARY:
The primary efficacy objective of this study is to establish the effect of burosumab treatment compared with placebo on increasing serum phosphorus levels in adults with XLH.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 - 65 years, inclusive
2. Diagnosis of XLH supported by classic clinical features of adult XLH (such as short stature or bowed legs) and at least ONE of the following at Screening:

   * Documented phosphate-regulating gene with homologies to endopeptidases on the X chromosome (PHEX) mutation in the patient or a directly related family member with appropriate X-linked inheritance
   * Serum intact FGF23 (iFGF23) level > 30 pg/mL by Kainos assay
3. Biochemical findings consistent with XLH at Screening Visit 2 following overnight fasting (min. 8 hours):

   * Serum phosphorus < 2.5 mg/dL
   * TmP/GFR of < 2.5 mg/dL
4. Presence of skeletal pain attributed to XLH/osteomalacia, as defined by a score of ≥ 4 on Brief Pain Inventory (BPI) Questions 3 (Worst Pain) at Screening Visit 1. (Skeletal pain that, in the opinion of the investigator, is attributed solely to causes other than XLH/osteomalacia-for example, back or joint pain in the presence of severe osteoarthritis by radiograph in that anatomical location-in the absence of any skeletal pain likely attributed to XLH/osteomalacia should not be considered for eligibility)
5. Estimated glomerular filtration rate (eGFR) ≥ 60 mL/min (using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation) or eGFR of 45 60 mL/min at Screening Visit 2 with confirmation that the renal insufficiency is not due to nephrocalcinosis
6. If taking chronic pain medications (including narcotic pain medications/opioids), must be on a stable regimen for at least 21 days prior to Screening Visit 1, and be willing to maintain medications at the same stable dose(s) and schedule throughout the Placebo-controlled Treatment Period of the study. The dose must not exceed 60 mg oral morphine equivalents/day
7. Provide written informed consent or if a minor, provide written consent and have a legally authorized representative willing and able to provide written informed consent, after the nature of the study has been explained, and prior to any research-related procedures
8. Willing to provide access to prior medical records for the collection of biochemical and radiographic data and disease history
9. Females of child-bearing potential must have a negative urine pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not to be of childbearing potential include those who have been in menopause for at least two years prior to Screening, or have had tubal ligation at least one year prior to Screening, or have had a total hysterectomy or bilateral salpingo-oophorectomy
10. Participants of child-bearing potential or with partners of child-bearing potential who have not undergone a bilateral salpingo-oophorectomy and are sexually active must consent to use an effective method of contraception as determined by the site investigator (i.e. oral hormonal contraceptives, patch hormonal contraceptives, vaginal ring, intrauterine device, physical double-barrier methods, surgical hysterectomy, vasectomy, tubal ligation, or true abstinence) from the period following the signing of the informed consent through 12 weeks after last dose of study drug
11. Must, in the opinion of the investigator, be willing and able to complete all aspects of the study, adhere to the study visit schedule and comply with the assessments
12. Must have completed at least 4 of 7 days of the patient diaries before the Baseline visit.

Exclusion Criteria:

1. Use of a pharmacologic vitamin D metabolite or analog (calcitriol, doxercalciferol, and paricalcitol) within 14 days prior to Screening Visit 2
2. Use of oral phosphate within 14 days prior to Screening Visit 2
3. Use of aluminum hydroxide antacids, acetazolamides, and thiazides within 7 days prior to Screening Visit 2
4. Chronic use of systemic corticosteroids defined as more than 10 days in the previous 2 months
5. Corrected serum calcium level ≥ 10.8 mg/dL (2.7 mmol/L) at Screening Visit 2
6. Serum intact parathyroid hormone (iPTH) ≥ 2.5 upper limit of normal (ULN) at Screening Visit 1
7. Use of medication to suppress parathyroid hormone (PTH) (cinacalcet for example) within 60 days prior to Screening Visit 1
8. Use of oral bisphosphonates for 6 months or more in the 2 years prior to Screening Visit 1
9. Use of denosumab in the 6 months prior to Screening Visit 1
10. Use of teriparatide in the 2 months prior to Screening Visit 1
11. Planned or recommended orthopedic surgery within the first 24 weeks of the clinical trial period
12. History of traumatic fracture or orthopedic surgery within 6 months prior to Screening Visit 1
13. Use of KRN23, or any other therapeutic monoclonal antibody within 90 days prior to Screening Visit 1
14. Use of any investigational product or investigational medical device within 30 days prior to Screening Visit 1, or requirement for any investigational agent prior to completion of all scheduled study assessments.

    OR, in Japan, use of any investigational product or investigational medical device within 4 months prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
15. Pregnant or breastfeeding at Screening /Baseline or planning to become pregnant (self or partner) at any time during the study
16. Unable or unwilling to withhold prohibited medications throughout the study
17. Presence or history of any hypersensitivity, allergic or anaphylactic reactions to any monoclonal antibody or KRN23 excipients that, in the judgment of the investigator, places the subject at increased risk for adverse effects.
18. Prior history of positive test for human immunodeficiency virus antibody, hepatitis B surface antigen, and/or hepatitis C antibody
19. History of recurrent infection or predisposition to infection, or of known immunodeficiency
20. Presence of malignant neoplasm (except basal cell carcinoma)
21. Presence of a concurrent disease or condition that would interfere with study participation or affect safety
22. Presence or history of any condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-10-22 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (25):
- United States (8):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California-San Francisco Medical Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Indiana University Department of Medicine, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Houston Methodist Hospital, Houston, Texas
- France (3):
  - CHU de Bicêtre, Service d'Endocrinologie et des Maladies de la Reproduction, Le Kremlin-Bicêtre
  - Hôpital Lariboisière, Dept. of Rheumatology, Paris
  - CHU Paris Centre-Hôpital Cochin, Paris
- St. Vincent's University Hospital, Dublin, Ireland
- Azienda Ospedaliero Universitaria Careggi - Neurofarba, Florence, Italy
- Japan (5):
  - Okayama Saiseikai General Hospital, Okayama
  - Osaka City University Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Toranomon Hospital, Tokyo
  - The University of Tokyo Hospital, Tokyo
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- United Kingdom (5):
  - University of Edinburgh Edinburgh Clinical Trials Unit (ECTU) - Western General Hospital, Edinburgh
  - Univeristy College of London Hospital, London
  - University of Oxford, Oxford
  - Northern General Hospital, Metabolic Bone Centre (Sorby Wing), Sheffield
  - Royal National Orthopaedic Hospital, Stanmore

REFERENCES:
- [Result] Insogna KL, Briot K, Imel EA, Kamenicky P, Ruppe MD, Portale AA, Weber T, Pitukcheewanont P, Cheong HI, Jan de Beur S, Imanishi Y, Ito N, Lachmann RH, Tanaka H, Perwad F, Zhang L, Chen CY, Theodore-Oklota C, Mealiffe M, San Martin J, Carpenter TO; AXLES 1 Investigators. A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial Evaluating the Efficacy of Burosumab, an Anti-FGF23 Antibody, in Adults With X-Linked Hypophosphatemia: Week 24 Primary Analysis. J Bone Miner Res. 2018 Aug;33(8):1383-1393. doi: 10.1002/jbmr.3475. Epub 2018 Jun 26. PMID 29947083
- [Result] Portale AA, Carpenter TO, Brandi ML, Briot K, Cheong HI, Cohen-Solal M, Crowley R, Jan De Beur S, Eastell R, Imanishi Y, Imel EA, Ing S, Ito N, Javaid M, Kamenicky P, Keen R, Kubota T, Lachmann R, Perwad F, Pitukcheewanont P, Ralston SH, Takeuchi Y, Tanaka H, Weber TJ, Yoo HW, Zhang L, Theodore-Oklota C, Mealiffe M, San Martin J, Insogna K. Continued Beneficial Effects of Burosumab in Adults with X-Linked Hypophosphatemia: Results from a 24-Week Treatment Continuation Period After a 24-Week Double-Blind Placebo-Controlled Period. Calcif Tissue Int. 2019 Sep;105(3):271-284. doi: 10.1007/s00223-019-00568-3. Epub 2019 Jun 4. PMID 31165191
- [Derived] Kamenicky P, Briot K, Brandi ML, Cohen-Solal M, Crowley RK, Keen R, Kolta S, Lachmann RH, Lecoq AL, Ralston SH, Walsh JS, Rylands AJ, Williams A, Sun W, Nixon A, Nixon M, Javaid MK. Benefit of burosumab in adults with X-linked hypophosphataemia (XLH) is maintained with long-term treatment. RMD Open. 2023 Feb;9(1):e002676. doi: 10.1136/rmdopen-2022-002676. PMID 36854566
- [Derived] Brandi ML, Jan de Beur S, Briot K, Carpenter T, Cheong HI, Cohen-Solal M, Crowley RK, Eastell R, Imanishi Y, Imel EA, Ing SW, Insogna K, Ito N, Javaid K, Kamenicky P, Keen R, Kubota T, Lachmann RH, Perwad F, Pitukcheewanont P, Portale A, Ralston SH, Tanaka H, Weber TJ, Yoo HW, Sun W, Williams A, Nixon A, Takeuchi Y. Efficacy of Burosumab in Adults with X-linked Hypophosphatemia (XLH): A Post Hoc Subgroup Analysis of a Randomized Double-Blind Placebo-Controlled Phase 3 Study. Calcif Tissue Int. 2022 Oct;111(4):409-418. doi: 10.1007/s00223-022-01006-7. Epub 2022 Aug 4. PMID 35927518
- [Derived] Briot K, Portale AA, Brandi ML, Carpenter TO, Cheong HI, Cohen-Solal M, Crowley RK, Eastell R, Imanishi Y, Ing S, Insogna K, Ito N, Jan de Beur S, Javaid MK, Kamenicky P, Keen R, Kubota T, Lachmann RH, Perwad F, Pitukcheewanont P, Ralston SH, Takeuchi Y, Tanaka H, Weber TJ, Yoo HW, Nixon A, Nixon M, Sun W, Williams A, Imel EA. Burosumab treatment in adults with X-linked hypophosphataemia: 96-week patient-reported outcomes and ambulatory function from a randomised phase 3 trial and open-label extension. RMD Open. 2021 Sep;7(3):e001714. doi: 10.1136/rmdopen-2021-001714. PMID 34548383

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subcutaneous (SC) injection of placebo every 4 weeks (Q4W) for 24 weeks (Double-blind Placebo-controlled Treatment Period), SC injection of burosumab 1 mg/kg Q4W for 24 weeks (Open-label Treatment Continuation Period), SC injection of burosumab 1 mg/kg Q4W for 48 weeks (Open-label Treatment Extension Period I), and SC injection of burosumab 1 mg/kg Q4W up to 53 weeks (Open-label Treatment Extension Period II).
- Burosumab 1 mg/kg: SC injection of 1.0 mg/kg burosumab Q4W for 24 weeks (double-blind placebo-controlled Treatment Period), SC injection of burosumab 1 mg/kg Q4W for 24 weeks (open-label Treatment Continuation Period), SC injection of burosumab 1 mg/kg Q4W for 48 weeks (open-label Treatment Extension Period I), and SC injection of burosumab 1 mg/kg Q4W up to 53 weeks (open-label Treatment Extension Period II).
Period: Double-Blind (Placebo-Controlled) Period
Arm/Group | Placebo | Burosumab 1 mg/kg
Started | 66 | 68
Completed | 66 | 67
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Open-label Treatment Continuation Period
Arm/Group | Placebo | Burosumab 1 mg/kg
Started | 66 | 67
Completed | 63 | 63
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other, Not Specified | 3 | 3
Period: Open-Label Treatment Extension Period I
Arm/Group | Placebo | Burosumab 1 mg/kg
Started | 63 | 63
Completed | 60 | 59
Not Completed | 3 | 4
Not completed — Death | 0 | 1
Not completed — Other, Not Specified | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Open-Label Treatment Extension Period II
Arm/Group | Placebo | Burosumab 1 mg/kg
Started | 52 | 49
Completed | 51 | 49
Not Completed | 1 | 0
Not completed — Other, Not Specified | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo SC Q4W through Week 24
- Burosumab: Burosumab 1 mg/kg SC Q4W
- Total: Total of all reporting groups
Arm/Group | Placebo | Burosumab | Total
Number analyzed (Participants) | 66 | 68 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.65 (12.756) | 41.29 (11.582) | 39.99 (12.201)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 44 | 87
  Male | 23 | 24 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 61 | 61 | 122
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 9 | 12 | 21
  Black or African American | 3 | 0 | 3
  White | 53 | 55 | 108
  Other, Not Specified | 1 | 1 | 2
Brief Pain Inventory (BPI) Worst Pain Score [Mean (Standard Deviation); unit: score on a scale] — The BPI evaluates the condition of all pain over the previous 24 hours. Question 3 of the short-form BPI (BPI-Q3) asks participants to rate their pain at its worst in the last 24 hours on a scale of 0 (no pain) to 10 (pain as bad as you can imagine). The baseline BPI Worst Pain is defined as the mean of the BPI Worst Pain for 8 days including the 7 days of diary scores prior to baseline visit and the baseline visit score.
  score on a scale | 6.54 (1.433) | 6.81 (1.308) | 6.68 (1.372)
BPI Pain Severity Score [Mean (Standard Deviation); unit: score on a scale] — The BPI evaluates the condition of all pain over the previous 24 hours. Two dimensions are measured: pain severity (worst, least, average, and now) and the impact of pain on functioning (pain interference with general activity, walking, work, mood, enjoyment of life, relations with others, and sleep). The severity of pain in the last 24 hours is rated on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
  score on a scale | 4.92 (1.547) | 5.18 (1.531) | 5.05 (1.539)
BPI Pain Interference Score [Mean (Standard Deviation); unit: score on a scale] — The BPI evaluates the condition of all pain over the previous 24 hours. Two dimensions are measured: pain severity (worst, least, average, and now) and the impact of pain on functioning (pain interference with general activity, walking, work, mood, enjoyment of life, relations with others, and sleep). Pain interference in the last 24 hours is rated on a scale of 0 (does not interfere) to 10 (completely interferes).
  score on a scale | 4.76 (2.174) | 5.23 (2.237) | 5.00 (2.210)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Score [Mean (Standard Deviation); unit: score on a scale] — The WOMAC is a 24-item participant-reported questionnaire with two domains, Stiffness (2 questions) and Physical Function (17 questions) over the previous 48 hours. The WOMAC is administered in a 5-point Likert-scale format using descriptors of none, mild, moderate, severe, and extreme corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse stiffness and functional limitations. Scores are normalized to a 0-100 metric where 0 was the best health state and 100 the worst.
  score on a scale | 61.36 (20.770) | 64.71 (20.253) | 63.06 (20.500)
WOMAC Physical Function Score [Mean (Standard Deviation); unit: score on a scale] — The WOMAC is a 24-item participant-reported questionnaire with two domains, Stiffness (2 questions) and Physical Function (17 questions) over the previous 48 hours. The WOMAC is administered in a 5-point Likert-scale format using descriptors of none, mild, moderate, severe, and extreme corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse stiffness and functional limitations. Scores are normalized to a 0-100 metric where 0 was the best health state and 100 the worst.
  score on a scale | 43.89 (19.938) | 50.79 (19.660) | 47.40 (20.024)
Brief Fatigue Inventory (BFI) Worst Fatigue Score [Mean (Standard Deviation); unit: score on a scale] — The BFI is a self-reported questionnaire consisting of 9 items related to fatigue rated on a 0 to 10 numerical scale with a recall period of 24 hours. Two dimensions are measured: fatigue severity and the interference of fatigue on daily life (activity, mood, walking ability, work, relations with others, and enjoyment of life). Participants are asked to rate their worst fatigue over the past 24 hours from 0 (no fatigue) to 10 (as bad a you can imagine).
  score on a scale | 6.74 (1.526) | 6.94 (1.657) | 6.84 (1.591)
BFI Global Fatigue Score [Mean (Standard Deviation); unit: score on a scale] — The BFI is a self-reported questionnaire consisting of 9 items related to fatigue that are rated on a numerical scale with a recall period of 24 hours. Two dimensions are measured: fatigue severity and the interference of fatigue on daily life (activity, mood, walking ability, work, relations with others, and enjoyment of life). BFI Global Fatigue score was calculated by averaging all 9 items on the BFI. Global scores range from 0 to 10, with higher score indicating worse fatigue severity and interference.
  score on a scale | 4.86 (1.932) | 5.37 (2.044) | 5.12 (1.999)
Serum Procollagen Type 1 N- Propeptide (P1NP) [Mean (Standard Deviation); unit: ng/mL] — Population: participants with a baseline assessment
  ng/mL
    number analyzed (Participants) | 66 | 67 | 133
    (all) | 87.6 (53.41) | 87.5 (53.60) | 87.6 (53.30)
Serum Carboxy-Terminal Cross-Linked Telopeptide of Type I Collagen (CTx) [Mean (Standard Deviation); unit: pg/mL] — Population: participants with a baseline assessment
  pg/mL
    number analyzed (Participants) | 66 | 67 | 133
    (all) | 719.2 (419.24) | 718.4 (413.71) | 718.8 (414.89)
Serum Bone-Specific Alkaline Phosphatase (BALP) [Mean (Standard Deviation); unit: μg/L] — Population: participants with a baseline assessment
  μg/L
    number analyzed (Participants) | 66 | 66 | 132
    (all) | 24.6 (17.30) | 25.1 (21.55) | 24.9 (19.47)
Serum Phosphorus [Mean (Standard Deviation); unit: mmol/L] | 0.617 (0.1001) | 0.653 (0.1072) | 0.635 (0.1050)
Serum 1, 25 (OH)2 D [Mean (Standard Deviation); unit: pg/mL] — Population: participants with a baseline assessment
  pg/mL
    number analyzed (Participants) | 64 | 66 | 130
    (all) | 33.5 (15.61) | 32.4 (12.96) | 33.0 (14.28)
24-Hour Urinary Phosphorus [Mean (Standard Deviation); unit: g/24 hour] — Population: participants with a baseline assessment
  g/24 hour
    number analyzed (Participants) | 65 | 68 | 133
    (all) | 0.81 (0.262) | 0.72 (0.241) | 0.77 (0.255)
Ratio of Renal Tubular Maximum Reabsorption Rate of Phosphate to Glomerular Filtration Rate(TmP/GFR) [Mean (Standard Deviation); unit: mg/dL] — Population: participants with a baseline assessment
  mg/dL
    number analyzed (Participants) | 64 | 66 | 130
    (all) | 1.598 (0.3693) | 1.678 (0.4004) | 1.639 (0.3860)
Tubular Reabsorption of Phosphate (TRP) [Mean (Standard Deviation); unit: fraction of phosphate reabsorbed] — Population: participants with a baseline assessment
  fraction of phosphate reabsorbed
    number analyzed (Participants) | 64 | 67 | 131
    (all) | 0.812 (0.0842) | 0.807 (0.0832) | 0.810 (0.0834)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Mean Serum Phosphorus Levels Above the LLN (2.5 mg/dL [0.81 mmol/L]) at the Mid-Point of the Dose Interval, as Averaged Across Dose Cycles Between Baseline and Week 24
Time Frame: Baseline through Week 24
Population: Primary Analysis Set: all randomized participants who received at least 1 dose of study drug during the Placebo-Controlled Treatment Period.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Burosumab
Number analyzed (Participants) | 66 | 68
percentage of participants | 7.6 [3.3 to 16.5] | 92.6 [83.9 to 96.8]
Statistical Analysis 1: Comparison: Placebo vs Burosumab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — From Cochran-Mantel-Haenszel (CMH) testing for association between achieving mean serum phosphorus levels above lower limit of normal (LLN) and treatment group, adjusting for stratification of Brief Pain Inventory (BPI) Average Pain and region

2. Secondary Outcome: Change From Baseline to Week 24 in Brief Pain Inventory (BPI) Question 3 (Q3; Worst Pain in Past 24 Hours) Score
Description: The BPI evaluates the condition of all pain over the previous 24 hours. Two dimensions are measured: pain severity (worst, least, average, and now) and the impact of pain on functioning (pain interference with general activity, walking, work, mood, enjoyment of life, relations with others, and sleep). Question 3 of the short-form BPI (BPI-Q3) asks subjects to rate their pain at its worst in the last 24 hours on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
  From the generalized estimating equation (GEE) model, which includes the change from Baseline for the endpoint of interest as the dependent variable; region, visit, treatment, actual randomization stratification (not included for analysis of BPI Worst Pain), and visit by treatment as fixed factors; and Baseline value for the endpoint of interest as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Burosumab
Number analyzed (Participants) | 66 | 68
score on a scale | -0.32 (0.222) | -0.79 (0.211)
Statistical Analysis 1: Comparison: Placebo vs Burosumab; Test type: Superiority; p = 0.0919, GEE model — Prespecified significance level for test after Hochberg adjustment: 0.05; Least squares (LS) mean difference = -0.46, 95% CI 2-sided [-1.00 to 0.08], Standard Error of Mean 0.275

3. Secondary Outcome: Change From Baseline to Week 24 in the Western Ontario and McMaster University Osteoarthritis Index (WOMAC) Stiffness Score
Description: The WOMAC is a 24-item participant-reported questionnaire with two domains, Stiffness (2 questions) and Physical Function (17 questions) over the previous 48 hours. The WOMAC is administered in a 5-point Likert-scale format using descriptors of none, mild, moderate, severe, and extreme corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse stiffness and functional limitations. Scores are normalized to a 0-100 metric where 0 was the best health state and 100 the worst.
  The GEE estimates are from the GEE model which includes the change from baseline for WOMAC Stiffness as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of WOMAC Stiffness as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Burosumab
Number analyzed (Participants) | 66 | 68
score on a scale | 0.46 (3.139) | -7.85 (3.034)
Statistical Analysis 1: Comparison: Placebo vs Burosumab; Test type: Superiority; p = 0.0106, GEE model — Prespecified significance level for test after Hochberg adjustment: 0.0167; LS mean difference = -8.31, 95% CI 2-sided [-14.68 to -1.94], Standard Error of Mean 3.251

4. Secondary Outcome: Change From Baseline to Week 24 in the WOMAC Physical Function Score
Description: The WOMAC is a 24-item participant-reported questionnaire with two domains, Stiffness (2 questions) and Physical Function (17 questions) over the previous 48 hours. The WOMAC is administered in a 5-point Likert-scale format using descriptors of none, mild, moderate, severe, and extreme corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse stiffness and functional limitations. Scores are normalized to a 0-100 metric where 0 was the best health state and 100 the worst.
  The GEE Estimates are from the GEE model which includes the change from baseline for WOMAC Physical Function as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of WOMAC Physical Function as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Burosumab
Number analyzed (Participants) | 66 | 68
score on a scale | 1.79 (2.722) | -3.11 (2.553)
Statistical Analysis 1: Comparison: Placebo vs Burosumab; Test type: Superiority; p = 0.0478, GEE model — Prespecified significance level for test after Hochberg adjustment: 0.025; LS mean difference = -4.9, 95% CI 2-sided [-9.76 to -0.05], Standard Error of Mean 2.479

5. Secondary Outcome: Change From Baseline Over Time in BPI Worst Pain Score
Description: Change from baseline to post-baseline visits in BPI-Q3 (Worst Pain) score as averaged from daily diary scores recorded over 1 week and the study visit score. The BPI evaluates the condition of all pain over the previous 24 hours. Two dimensions are measured: pain severity (worst, least, average, and now) and the impact of pain on functioning (pain interference with general activity, walking, work, mood, enjoyment of life, relations with others, and sleep). Question 3 of the short-form BPI (BPI-Q3) asks subjects to rate their pain at its worst in the last 24 hours on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
  The GEE Estimates are from the GEE model which includes the change from baseline for BPI worst pain as the dependent variable, region, visit, treatment and visit by treatment as fixed factors, and baseline of BPI Worst Pain as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96
Population: Primary Analysis Set: all randomized participants who received at least 1 dose of study drug during the Placebo-Controlled Treatment Period. Participants with an assessment at given time point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 68
score on a scale
  Change at Week 12 | -0.37 (0.216) | -0.62 (0.208)
  Change at Week 24: number analyzed (Participants) | 65 | 67
  Change at Week 24 | -0.31 (0.242) | -0.77 (0.228)
  Change at Week 36: number analyzed (Participants) | 65 | 65
  Change at Week 36 | -1.25 (0.234) | -0.95 (0.228)
  Change at Week 48: number analyzed (Participants) | 66 | 66
  Change at Week 48 | -1.49 (0.243) | -1.05 (0.230)
  Change at Week 72: number analyzed (Participants) | 60 | 59
  Change at Week 72 | -1.28 (0.283) | -1.21 (0.316)
  Change at Week 96: number analyzed (Participants) | 59 | 59
  Change at Week 96 | -0.99 (0.265) | -1.48 (0.299)

6. Secondary Outcome: Change From Baseline Over Time in BPI Pain Severity Score
Description: Change from baseline to post-baseline visits in BPI pain severity score as averaged from daily diary scores recorded over 1 week and the study visit score. The BPI evaluates the condition of all pain over the previous 24 hours. Two dimensions are measured: pain severity (worst, least, average, and now) and the impact of pain on functioning (pain interference with general activity, walking, work, mood, enjoyment of life, relations with others, and sleep). The severity of pain in the last 24 hours is rated on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
  The GEE Estimates are from the GEE model which includes the change from baseline for each BPI endpoint as the dependent variable, region, visit, treatment, and visit by treatment as fixed factors, and baseline of each BPI endpoint as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 68
score on a scale
  Change at Week 12 | -0.32 (0.166) | -0.43 (0.163)
  Change at Week 24: number analyzed (Participants) | 65 | 67
  Change at Week 24 | -0.10 (0.211) | -0.53 (0.172)
  Change at Week 36: number analyzed (Participants) | 65 | 65
  Change at Week 36 | -0.97 (0.214) | -0.62 (0.184)
  Change at Week 48: number analyzed (Participants) | 66 | 66
  Change at Week 48 | -1.13 (0.205) | -0.79 (0.162)
  Change at Week 72: number analyzed (Participants) | 60 | 59
  Change at Week 72 | -1.36 (0.216) | -1.24 (0.231)
  Change at Week 96: number analyzed (Participants) | 59 | 59
  Change at Week 96 | -1.18 (0.195) | -1.42 (0.229)

7. Secondary Outcome: Change From Baseline Over Time in BPI Pain Interference Score
Description: Change from baseline to post-baseline visits in BPI pain interference score as recorded on the day of the study visit. The BPI evaluates the condition of all pain over the previous 24 hours. Two dimensions are measured: pain severity (worst, least, average, and now) and the impact of pain on functioning (pain interference with general activity, walking, work, mood, enjoyment of life, relations with others, and sleep). Pain interference in the last 24 hours is rated on a scale of 0 (does not interfere) to 10 (completely interferes).
  The GEE Estimates are from the GEE model which includes the change from baseline for each BPI endpoint as the dependent variable, region, visit, treatment, and visit by treatment as fixed factors, and baseline of each BPI endpoint as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 68
score on a scale
  Change at Week 12 | -0.29 (0.215) | -0.51 (0.207)
  Change at Week 24: number analyzed (Participants) | 65 | 67
  Change at Week 24 | -0.28 (0.242) | -0.41 (0.207)
  Change at Week 36: number analyzed (Participants) | 65 | 65
  Change at Week 36 | -1.30 (0.260) | -0.79 (0.221)
  Change at Week 48: number analyzed (Participants) | 66 | 66
  Change at Week 48 | -1.28 (0.251) | -1.04 (0.235)
  Change at Week 72: number analyzed (Participants) | 60 | 60
  Change at Week 72 | -1.22 (0.247) | -1.24 (0.263)
  Change at Week 96: number analyzed (Participants) | 59 | 59
  Change at Week 96 | -1.08 (0.260) | -1.43 (0.234)

8. Secondary Outcome: Change From Baseline Over Time in WOMAC Stiffness Score
Description: as for outcome 3
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96, 120, 144
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 68
score on a scale
  Change at Week 12 | -1.24 (2.929) | -7.86 (3.622)
  Change at Week 24: number analyzed (Participants) | 65 | 67
  Change at Week 24 | 0.20 (3.289) | -8.01 (2.968)
  Change at Week 36: number analyzed (Participants) | 65 | 65
  Change at Week 36 | -13.50 (3.422) | -12.58 (3.411)
  Change at Week 48: number analyzed (Participants) | 66 | 66
  Change at Week 48 | -15.83 (3.488) | -16.63 (3.302)
  Change at Week 72: number analyzed (Participants) | 61 | 60
  Change at Week 72 | -18.02 (3.613) | -15.47 (3.111)
  Change at Week 96: number analyzed (Participants) | 59 | 59
  Change at Week 96 | -17.67 (3.737) | -15.32 (3.577)
  Change at Week 120: number analyzed (Participants) | 49 | 46
  Change at Week 120 | -19.23 (3.404) | -20.57 (3.371)
  Change at Week 144: number analyzed (Participants) | 9 | 12
  Change at Week 144 | -30.64 (4.407) | -25.88 (4.501)

9. Secondary Outcome: Change From Baseline Over Time in WOMAC Physical Function Score
Description: as for outcome 3
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96, 120, 144
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 68
score on a scale
  Change at Week 12 | -1.40 (2.418) | -3.96 (1.787)
  Change at Week 24: number analyzed (Participants) | 65 | 66
  Change at Week 24 | 1.14 (2.531) | -3.45 (2.193)
  Change at Week 36: number analyzed (Participants) | 63 | 65
  Change at Week 36 | -5.47 (2.694) | -7.14 (2.133)
  Change at Week 48: number analyzed (Participants) | 66 | 66
  Change at Week 48 | -7.15 (2.801) | -8.42 (2.057)
  Change at Week 72: number analyzed (Participants) | 61 | 60
  Change at Week 72 | -8.68 (2.835) | -8.66 (2.523)
  Change at Week 96: number analyzed (Participants) | 59 | 59
  Change at Week 96 | -8.41 (2.752) | -9.02 (2.270)
  Change at Week 120: number analyzed (Participants) | 49 | 46
  Change at Week 120 | -11.93 (2.685) | -11.98 (2.291)
  Change at Week 144: number analyzed (Participants) | 9 | 11
  Change at Week 144 | -19.49 (3.892) | -17.67 (4.061)

10. Secondary Outcome: Change From Baseline Over Time in BFI Worst Fatigue Score
Description: Change from baseline to post-baseline visits in Brief Fatigue Inventory Question 3 (Worst Fatigue in Past 24 Hours; BFI-Q3) as averaged from daily diary scores recorded over 1 week and the study visit score. The BFI is a self-reported questionnaire consisting of 9 items related to fatigue rated on a 0 to 10 numerical scale with a recall period of 24 hours. Two dimensions are measured: fatigue severity and the interference of fatigue on daily life (activity, mood, walking ability, work, relations with others, and enjoyment of life). Participants are asked to rate their worst fatigue over the past 24 hours from 0 (no fatigue) to 10 (as bad a you can imagine).
  The GEE Estimates are from the GEE model which includes the change from baseline for each BFI endpoint as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of each BFI endpoint as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 68
score on a scale
  Change at Week 12 | -0.53 (0.266) | -0.44 (0.261)
  Change at Week 24: number analyzed (Participants) | 65 | 67
  Change at Week 24 | -0.45 (0.298) | -0.65 (0.280)
  Change at Week 36: number analyzed (Participants) | 65 | 65
  Change at Week 36 | -1.23 (0.305) | -0.90 (0.271)
  Change at Week 48: number analyzed (Participants) | 66 | 66
  Change at Week 48 | -1.21 (0.317) | -0.99 (0.295)
  Change at Week 72: number analyzed (Participants) | 60 | 60
  Change at Week 72 | -0.79 (0.352) | -0.58 (0.309)
  Change at Week 96: number analyzed (Participants) | 59 | 58
  Change at Week 96 | -0.82 (0.362) | -0.75 (0.306)

11. Secondary Outcome: Change From Baseline Over Time in BFI Global Fatigue Score
Description: Change from baseline to post-baseline visits in BFI global fatigue score, calculated by averaging all 9 BFI items as recorded on the day of the study visit. The BFI is a self-reported questionnaire consisting of 9 items related to fatigue that are rated on a numerical scale with a recall period of 24 hours. Two dimensions are measured: fatigue severity and the interference of fatigue on daily life (activity, mood, walking ability, work, relations with others, and enjoyment of life). BFI Global Fatigue score was calculated by averaging all 9 items on the BFI. Global scores range from 0 to 10, with higher score indicating worse fatigue severity and interference.
  The GEE Estimates are from the GEE model which includes the change from baseline for each BFI endpoint as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of each BFI endpoint as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: SC injection of placebo Q4W for 24 weeks (Double-blind Placebo-controlled Treatment Period), SC injection of burosumab 1 mg/kg Q4W for 24 weeks (Open-label Treatment Continuation Period), SC injection of burosumab 1 mg/kg Q4W for 48 weeks (Open-label Treatment Extension Period I), and SC injection of burosumab 1 mg/kg Q4W up to 53 weeks (Open-label Treatment Extension Period II).
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 68
score on a scale
  Change at Week 12 | -0.14 (0.262) | -0.18 (0.261)
  Change at Week 24: number analyzed (Participants) | 65 | 67
  Change at Week 24 | -0.08 (0.292) | 0.05 (0.261)
  Change at Week 36: number analyzed (Participants) | 65 | 65
  Change at Week 36 | -0.69 (0.315) | -0.54 (0.283)
  Change at Week 48: number analyzed (Participants) | 66 | 66
  Change at Week 48 | -0.75 (0.303) | -0.45 (0.275)
  Change at Week 72: number analyzed (Participants) | 60 | 60
  Change at Week 72 | -0.72 (0.304) | -0.78 (0.266)
  Change at Week 96: number analyzed (Participants) | 59 | 58
  Change at Week 96 | -0.86 (0.291) | -0.80 (0.285)

12. Secondary Outcome: Change From Baseline Over Time in Biochemical Marker of Bone Remodeling Procollagen Type 1 N-Propeptide (P1NP)
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 67
ng/mL
  Change at Week 12 | -1.86 (5.958) | 96.22 (14.264)
  Change at Week 24: number analyzed (Participants) | 65 | 66
  Change at Week 24 | 2.95 (6.423) | 63.50 (7.239)
  Change at Week 36: number analyzed (Participants) | 65 | 64
  Change at Week 36 | 100.00 (10.562) | 49.71 (6.786)
  Change at Week 48: number analyzed (Participants) | 66 | 63
  Change at Week 48 | 85.12 (11.037) | 40.07 (7.292)
  Change at Week 72: number analyzed (Participants) | 60 | 59
  Change at Week 72 | 48.98 (7.286) | 18.04 (9.186)
  Change at Week 96: number analyzed (Participants) | 59 | 59
  Change at Week 96 | 22.98 (7.075) | 12.48 (8.661)

13. Secondary Outcome: Percent Change From Baseline Over Time in Biochemical Marker of Bone Remodeling P1NP
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 67
percentage change
  Change at Week 12 | 2.30 (6.318) | 91.78 (10.787)
  Change at Week 24: number analyzed (Participants) | 65 | 66
  Change at Week 24 | 7.83 (7.076) | 72.43 (8.519)
  Change at Week 36: number analyzed (Participants) | 65 | 64
  Change at Week 36 | 116.39 (9.726) | 63.58 (8.562)
  Change a Week 48: number analyzed (Participants) | 66 | 63
  Change a Week 48 | 99.10 (11.442) | 56.51 (8.771)
  Change at Week 72: number analyzed (Participants) | 60 | 59
  Change at Week 72 | 72.56 (10.055) | 38.82 (10.225)
  Change at Week 96: number analyzed (Participants) | 59 | 59
  Change at Week 96 | 41.62 (8.163) | 31.04 (8.126)

14. Secondary Outcome: Change From Baseline Over Time in Biochemical Marker of Bone Remodeling Carboxy-Terminal Cross-Linked Telopeptide of Type I Collagen (CTx)
Description: The GEE Estimates are from the GEE model which includes the change from baseline for CTx as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of CTx as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 67
pg/mL
  Change at Week 12 | 26.96 (35.689) | 322.09 (56.924)
  Change at Week 24: number analyzed (Participants) | 64 | 66
  Change at Week 24 | -4.20 (34.835) | 184.56 (39.213)
  Change at Week 36: number analyzed (Participants) | 65 | 63
  Change at Week 36 | 350.89 (53.131) | 193.50 (39.461)
  Change at Week 48: number analyzed (Participants) | 66 | 63
  Change at Week 48 | 310.67 (45.003) | 138.61 (37.886)
  Change at Week 72: number analyzed (Participants) | 60 | 59
  Change at Week 72 | 178.03 (42.702) | 51.59 (42.863)
  Change at Week 96: number analyzed (Participants) | 59 | 59
  Change at Week 96 | 79.04 (45.622) | 10.84 (40.761)

15. Secondary Outcome: Percent Change From Baseline Over Time in Biochemical Marker of Bone Remodeling CTx
Description: The GEE Estimates are from the GEE model which includes the percent change from baseline for CTx as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of CTx as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 67
percentage change
  Change at Week 12 | 9.64 (5.671) | 45.40 (7.267)
  Change at Week 24: number analyzed (Participants) | 64 | 66
  Change at Week 24 | 4.75 (5.280) | 32.48 (6.414)
  Change at Week 36: number analyzed (Participants) | 65 | 63
  Change at Week 36 | 61.31 (10.653) | 34.07 (6.250)
  Change at Week 48: number analyzed (Participants) | 66 | 63
  Change at Week 48 | 50.35 (6.464) | 28.33 (5.354)
  Change at Week 72: number analyzed (Participants) | 60 | 59
  Change at Week 72 | 34.78 (7.007) | 17.09 (5.957)
  Change at Week 96: number analyzed (Participants) | 59 | 59
  Change at Week 96 | 27.38 (7.783) | 13.47 (5.952)

16. Secondary Outcome: Change From Baseline Over Time in Biochemical Marker of Bone Remodeling Bone-Specific Alkaline Phosphatase (BALP)
Description: The GEE Estimates are from the GEE model which includes the change from baseline for BALP as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of BALP as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: μg/L
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 66
μg/L
  Change at Week 12 | -2.11 (1.529) | 6.52 (2.832)
  Change at Week 24: number analyzed (Participants) | 64 | 65
  Change at Week 24 | 1.03 (1.801) | 5.70 (2.038)
  Change at Week 36: number analyzed (Participants) | 65 | 63
  Change at Week 36 | 10.42 (2.017) | 4.46 (1.607)
  Change at Week 48: number analyzed (Participants) | 66 | 61
  Change at Week 48 | 6.69 (1.929) | 0.23 (1.830)
  Change at Week 72: number analyzed (Participants) | 61 | 58
  Change at Week 72 | -0.92 (1.779) | -3.39 (1.739)
  Change at Week 96: number analyzed (Participants) | 59 | 58
  Change at Week 96 | -2.49 (1.887) | -2.76 (1.640)

17. Secondary Outcome: Percent Change From Baseline Over Time in Biochemical Marker of Bone Remodeling BALP
Description: The GEE Estimates are from the GEE model which includes the percent change from baseline for BALP as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of Bone ALP as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 66
percentage change
  Change at Week 12 | 7.85 (9.867) | 30.29 (13.476)
  Change at Week 24: number analyzed (Participants) | 64 | 65
  Change at Week 24 | 27.56 (10.339) | 39.13 (10.902)
  Change at Week 36: number analyzed (Participants) | 65 | 63
  Change at Week 36 | 64.41 (11.669) | 43.13 (11.473)
  Change at Week 48: number analyzed (Participants) | 66 | 61
  Change at Week 48 | 50.65 (11.317) | 23.46 (10.041)
  Change at Week 72: number analyzed (Participants) | 61 | 58
  Change at Week 72 | 19.79 (11.755) | 14.40 (11.618)
  Change at Week 96: number analyzed (Participants) | 59 | 58
  Change at Week 96 | 16.46 (11.027) | 21.21 (9.688)

18. Secondary Outcome: Change From Baseline Over Time in Serum Phosphorus
Description: The GEE Estimates are from the GEE model which includes the change from baseline for serum phosphorus as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of serum phosphorus as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 10, 12, 14, 18, 20, 21, 22, 24, 26, 28, 34, 36, 46, 48, 60, 70, 72, 84, 94, 96, 108, 120, 132, 144
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 68
mmol/L
  Change at Week 1: number analyzed (Participants) | 60 | 61
  Change at Week 1 | -0.01 (0.024) | 0.44 (0.031)
  Change at Week 2: number analyzed (Participants) | 64 | 64
  Change at Week 2 | -0.03 (0.023) | 0.43 (0.032)
  Change at Week 4: number analyzed (Participants) | 65 | 67
  Change at Week 4 | -0.03 (0.022) | 0.27 (0.034)
  Change at Week 6: number analyzed (Participants) | 65 | 65
  Change at Week 6 | -0.00 (0.023) | 0.45 (0.036)
  Change at Week 10: number analyzed (Participants) | 64 | 64
  Change at Week 10 | 0.01 (0.022) | 0.37 (0.033)
  Change at Week 12: number analyzed (Participants) | 64 | 68
  Change at Week 12 | -0.01 (0.023) | 0.17 (0.032)
  Change at Week 14: number analyzed (Participants) | 66 | 65
  Change at Week 14 | 0.02 (0.022) | 0.32 (0.032)
  Change at Week 18: number analyzed (Participants) | 62 | 68
  Change at Week 18 | 0.02 (0.023) | 0.32 (0.031)
  Change at Week 20: number analyzed (Participants) | 65 | 65
  Change at Week 20 | -0.01 (0.023) | 0.18 (0.028)
  Change at Week 21: number analyzed (Participants) | 61 | 65
  Change at Week 21 | -0.00 (0.024) | 0.31 (0.033)
  Change at Week 22: number analyzed (Participants) | 65 | 64
  Change at Week 22 | -0.02 (0.022) | 0.25 (0.033)
  Change at Week 24 | -0.00 (0.023) | 0.13 (0.028)
  Change at Week 26: number analyzed (Participants) | 62 | 66
  Change at Week 26 | 0.47 (0.035) | 0.31 (0.032)
  Change at Week 28: number analyzed (Participants) | 66 | 67
  Change at Week 28 | 0.28 (0.028) | 0.18 (0.028)
  Change at Week 34: number analyzed (Participants) | 65 | 62
  Change at Week 34 | 0.36 (0.029) | 0.28 (0.031)
  Change at Week 36: number analyzed (Participants) | 66 | 64
  Change at Week 36 | 0.17 (0.026) | 0.13 (0.027)
  Change at Week 46: number analyzed (Participants) | 66 | 65
  Change at Week 46 | 0.31 (0.026) | 0.27 (0.030)
  Change at Week 48: number analyzed (Participants) | 66 | 64
  Change at Week 48 | 0.13 (0.027) | 0.11 (0.027)
  Change at Week 60: number analyzed (Participants) | 62 | 61
  Change at Week 60 | 0.14 (0.028) | 0.11 (0.028)
  Change at Week 70: number analyzed (Participants) | 55 | 57
  Change at Week 70 | 0.30 (0.029) | 0.30 (0.030)
  Change at Week 72: number analyzed (Participants) | 61 | 60
  Change at Week 72 | 0.13 (0.025) | 0.11 (0.027)
  Change at Week 84: number analyzed (Participants) | 60 | 59
  Change at Week 84 | 0.12 (0.025) | 0.14 (0.027)
  Change at Week 94: number analyzed (Participants) | 59 | 58
  Change at Week 94 | 0.25 (0.029) | 0.30 (0.029)
  Change at Week 96: number analyzed (Participants) | 60 | 59
  Change at Week 96 | 0.07 (0.026) | 0.13 (0.025)
  Change at Week 108: number analyzed (Participants) | 49 | 48
  Change at Week 108 | 0.11 (0.028) | 0.13 (0.031)
  Change at Week 120: number analyzed (Participants) | 44 | 41
  Change at Week 120 | 0.09 (0.027) | 0.13 (0.033)
  Change at Week 132: number analyzed (Participants) | 19 | 19
  Change at Week 132 | 0.12 (0.033) | 0.15 (0.036)
  Change at Week 144: number analyzed (Participants) | 2 | 0
  Change at Week 144 | 0.05 (0.064) |

19. Secondary Outcome: Percent Change From Baseline Over Time in Serum Phosphorus
Description: The GEE Estimates are from the GEE model which includes the percent change from baseline for serum phosphorus as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of serum phosphorus as a covariate, with compound symmetry covariance structure.
Time Frame: as for outcome 18
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 66 | 68
percentage change
  Change at Week 1: number analyzed (Participants) | 60 | 61
  Change at Week 1 | -1.11 (3.936) | 69.24 (4.762)
  Change at Week 2: number analyzed (Participants) | 64 | 64
  Change at Week 2 | -5.91 (3.969) | 69.39 (4.881)
  Change at Week 4: number analyzed (Participants) | 65 | 67
  Change at Week 4 | -4.84 (3.792) | 42.89 (5.325)
  Change at Week 6: number analyzed (Participants) | 65 | 65
  Change at Week 6 | -0.41 (3.951) | 72.96 (5.944)
  Change at Week 10: number analyzed (Participants) | 64 | 64
  Change at Week 10 | 2.40 (3.680) | 59.96 (5.356)
  Change at Week 12: number analyzed (Participants) | 64 | 68
  Change at Week 12 | -2.14 (3.798) | 29.50 (5.087)
  Change at Week 14: number analyzed (Participants) | 66 | 65
  Change at Week 14 | 3.58 (3.691) | 52.14 (5.194)
  Change at Week 18: number analyzed (Participants) | 62 | 68
  Change at Week 18 | 3.93 (3.857) | 53.22 (5.106)
  Change at Week 20: number analyzed (Participants) | 65 | 65
  Change at Week 20 | -1.81 (3.759) | 31.28 (4.472)
  Change at Week 21: number analyzed (Participants) | 61 | 65
  Change at Week 21 | 0.21 (4.011) | 50.59 (5.123)
  Change at Week 22: number analyzed (Participants) | 65 | 64
  Change at Week 22 | -3.42 (3.709) | 40.98 (5.196)
  Change at Week 24 | -0.61 (3.802) | 22.01 (4.523)
  Change at Week 26: number analyzed (Participants) | 62 | 66
  Change at Week 26 | 78.30 (5.993) | 51.51 (5.204)
  Change at Week 28: number analyzed (Participants) | 66 | 67
  Change at Week 28 | 46.07 (4.766) | 31.32 (4.415)
  Change at Week 34: number analyzed (Participants) | 65 | 62
  Change at Week 34 | 59.18 (4.959) | 45.83 (4.871)
  Change at Week 36: number analyzed (Participants) | 66 | 64
  Change at Week 36 | 28.03 (4.424) | 22.34 (4.256)
  Change at Week 46: number analyzed (Participants) | 66 | 65
  Change at Week 46 | 51.49 (4.380) | 45.39 (5.018)
  Change at Week 48: number analyzed (Participants) | 66 | 64
  Change at Week 48 | 21.58 (4.365) | 19.12 (4.190)
  Change at Week 60: number analyzed (Participants) | 62 | 61
  Change at Week 60 | 22.90 (4.338) | 19.60 (4.436)
  Change at Week 70: number analyzed (Participants) | 55 | 57
  Change at Week 70 | 50.22 (4.916) | 47.81 (4.768)
  Change at Week 72: number analyzed (Participants) | 61 | 60
  Change at Week 72 | 21.59 (4.155) | 19.45 (4.344)
  Change at Week 84: number analyzed (Participants) | 60 | 59
  Change at Week 84 | 21.47 (4.089) | 23.58 (4.200)
  Change at Week 94: number analyzed (Participants) | 59 | 58
  Change at Week 94 | 43.67 (4.834) | 49.36 (4.501)
  Change at Week 96: number analyzed (Participants) | 60 | 59
  Change at Week 96 | 12.97 (4.216) | 21.65 (3.854)
  Change at Week 108: number analyzed (Participants) | 49 | 48
  Change at Week 108 | 19.21 (4.665) | 23.39 (4.749)
  Change at Week 120: number analyzed (Participants) | 44 | 41
  Change at Week 120 | 15.13 (4.365) | 21.50 (5.268)
  Change at Week 132: number analyzed (Participants) | 19 | 19
  Change at Week 132 | 20.43 (5.362) | 25.34 (5.847)
  Change at Week 144: number analyzed (Participants) | 2 | 0
  Change at Week 144 | 5.49 (12.212) |

20. Secondary Outcome: Change From Baseline Over Time in Serum 1,25(OH)2D
Description: The GEE Estimates are from the GEE model which includes the change from baseline for 1,25(OH)2D as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of 1, 25 (OH)2 D as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 1, 2, 4, 20, 21, 22, 46, 48, 60, 70, 72, 84, 94, 96, 108, 120, 132, 144
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 64 | 66
pg/mL
  Change at Week 1: number analyzed (Participants) | 58 | 59
  Change at Week 1 | 2.04 (2.251) | 87.23 (5.500)
  Change at Week 2: number analyzed (Participants) | 63 | 65
  Change at Week 2 | 1.40 (2.113) | 58.20 (3.931)
  Change at Week 4: number analyzed (Participants) | 63 | 66
  Change at Week 4 | 2.61 (2.300) | 20.55 (2.828)
  Change at Week 20: number analyzed (Participants) | 64 | 63
  Change at Week 20 | 2.88 (2.163) | 8.11 (2.294)
  Change at Week 21: number analyzed (Participants) | 59 | 64
  Change at Week 21 | 3.09 (2.177) | 33.95 (3.019)
  Change at Week 22: number analyzed (Participants) | 64 | 65
  Change at Week 22 | 3.45 (2.289) | 26.10 (2.952)
  Change at Week 46: number analyzed (Participants) | 64 | 64
  Change at Week 46 | 25.23 (2.576) | 23.08 (3.243)
  Change at Week 48: number analyzed (Participants) | 64 | 63
  Change at Week 48 | 10.50 (2.418) | 7.24 (2.449)
  Change at Week 60: number analyzed (Participants) | 59 | 60
  Change at Week 60 | 9.29 (2.336) | 5.69 (2.583)
  Change at Week 70: number analyzed (Participants) | 54 | 60
  Change at Week 70 | 24.20 (2.529) | 18.82 (2.486)
  Change at Week 72: number analyzed (Participants) | 59 | 58
  Change at Week 72 | 7.12 (2.424) | 5.52 (2.607)
  Change at Week 84: number analyzed (Participants) | 58 | 57
  Change at Week 84 | 5.13 (2.388) | 1.16 (2.549)
  Change at Week 94: number analyzed (Participants) | 57 | 58
  Change at Week 94 | 18.96 (2.655) | 15.26 (2.502)
  Change at Week 96: number analyzed (Participants) | 56 | 58
  Change at Week 96 | 3.43 (2.348) | 1.95 (2.356)
  Change at Week 108: number analyzed (Participants) | 48 | 48
  Change at Week 108 | 4.76 (2.349) | 4.29 (2.672)
  Change at Week 120: number analyzed (Participants) | 43 | 42
  Change at Week 120 | 4.64 (2.496) | 5.37 (2.935)
  Change at Week 132: number analyzed (Participants) | 18 | 19
  Change at Week 132 | 4.08 (3.142) | 8.05 (4.227)
  Change at Week 144: number analyzed (Participants) | 2 | 0
  Change at Week 144 | -0.38 (4.677) |

21. Secondary Outcome: Percent Change From Baseline Over Time in Serum 1,25(OH)2D
Description: The GEE Estimates are from the GEE model which includes the percent change from baseline for 1,25(OH)2D as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of 1, 25 (OH)2 D as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 1, 2, 4, 20, 21, 22, 46, 48, 60, 70, 72, 84, 94, 96, 108, 120, 132, 144
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 64 | 66
percentage change
  Change at Week 1: number analyzed (Participants) | 58 | 59
  Change at Week 1 | 10.45 (13.041) | 310.72 (23.225)
  Change at Week 2: number analyzed (Participants) | 63 | 65
  Change at Week 2 | 10.53 (12.760) | 207.90 (16.728)
  Change at Week 4: number analyzed (Participants) | 63 | 66
  Change at Week 4 | 16.07 (12.810) | 76.22 (12.147)
  Change at Week 20: number analyzed (Participants) | 64 | 63
  Change at Week 20 | 21.36 (12.424) | 41.08 (11.943)
  Change at Week 21: number analyzed (Participants) | 59 | 64
  Change at Week 21 | 21.51 (12.825) | 131.76 (14.862)
  Change at Week 22: number analyzed (Participants) | 64 | 65
  Change at Week 22 | 21.07 (12.725) | 102.81 (14.619)
  Change at Week 46: number analyzed (Participants) | 64 | 64
  Change at Week 46 | 130.29 (22.718) | 96.63 (16.909)
  Change at Week 48: number analyzed (Participants) | 64 | 63
  Change at Week 48 | 70.09 (17.114) | 34.47 (12.903)
  Change at Week 60: number analyzed (Participants) | 59 | 60
  Change at Week 60 | 65.46 (13.083) | 32.32 (12.230)
  Change at Week 70: number analyzed (Participants) | 54 | 60
  Change at Week 70 | 123.58 (17.315) | 82.03 (12.604)
  Change at Week 72: number analyzed (Participants) | 59 | 58
  Change at Week 72 | 58.45 (13.957) | 31.14 (13.070)
  Change at Week 84: number analyzed (Participants) | 58 | 57
  Change at Week 84 | 55.67 (15.323) | 18.83 (12.801)
  Change at Week 94: number analyzed (Participants) | 57 | 58
  Change at Week 94 | 111.25 (21.970) | 71.30 (12.280)
  Change at Week 96: number analyzed (Participants) | 56 | 58
  Change at Week 96 | 50.17 (18.857) | 22.15 (10.487)
  Change at Week 108: number analyzed (Participants) | 48 | 48
  Change at Week 108 | 44.78 (14.219) | 29.16 (13.326)
  Change at Week 120: number analyzed (Participants) | 43 | 42
  Change at Week 120 | 58.37 (19.621) | 36.09 (13.089)
  Change at Week 132: number analyzed (Participants) | 18 | 19
  Change at Week 132 | 67.59 (35.770) | 42.55 (15.925)
  Change at Week 144: number analyzed (Participants) | 2 | 0
  Change at Week 144 | 22.65 (19.297) |

22. Secondary Outcome: Change From Baseline Over Time in 24-Hour Urinary Phosphorus
Description: The GEE Estimates are from the GEE model which includes the change from baseline for 24-Hour urinary phosphorus as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of urinary phosphorus as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Week 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: g/24 hour
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 65 | 67
g/24 hour
  Change at Week 12: number analyzed (Participants) | 63 | 63
  Change at Week 12 | 0.06 (0.052) | 0.05 (0.046)
  Change at Week 24 | 0.07 (0.065) | 0.05 (0.046)
  Change at Week 36: number analyzed (Participants) | 64 | 64
  Change at Week 36 | 0.04 (0.054) | 0.07 (0.045)
  Change at Week 48: number analyzed (Participants) | 63 | 63
  Change at Week 48 | 0.07 (0.060) | 0.13 (0.067)
  Change at Week 72: number analyzed (Participants) | 57 | 57
  Change at Week 72 | 0.08 (0.065) | 0.05 (0.052)
  Change at Week 96: number analyzed (Participants) | 58 | 59
  Change at Week 96 | 0.10 (0.075) | 0.10 (0.054)

23. Secondary Outcome: Percent Change From Baseline Over Time in 24-Hour Urinary Phosphorus
Description: The GEE Estimates are from the GEE model which includes the percent change from baseline for 24-hour urinary phosphorus as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of urinary phosphorus as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Week 12, 24, 36, 48, 72, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 65 | 67
percentage change
  Change at Week 12: number analyzed (Participants) | 63 | 63
  Change at Week 12 | 21.91 (11.844) | 21.40 (11.453)
  Change at Week 24 | 28.45 (15.518) | 20.35 (11.567)
  Change at Week 36: number analyzed (Participants) | 64 | 64
  Change at Week 36 | 18.19 (11.784) | 28.31 (12.173)
  Change at Week 48: number analyzed (Participants) | 63 | 63
  Change at Week 48 | 27.32 (14.328) | 37.50 (14.687)
  Change at Week 72: number analyzed (Participants) | 57 | 57
  Change at Week 72 | 29.53 (14.485) | 25.80 (15.476)
  Change at Week 96: number analyzed (Participants) | 58 | 59
  Change at Week 96 | 31.17 (17.248) | 30.64 (10.420)

24. Secondary Outcome: Change From Baseline Over Time in Ratio of Renal Tubular Maximum Reabsorption Rate of Phosphate to Glomerular Filtration Rate (TmP/GFR)
Description: The GEE Estimates are from the GEE model which includes the change from baseline for TmP/GFR as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of TmP/GFR as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 2, 4, 12, 22, 24, 48, 60, 72, 84, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 63 | 66
mg/dL
  Change at Week 2: number analyzed (Participants) | 60 | 60
  Change at Week 2 | -0.02 (0.072) | 1.60 (0.121)
  Change at Week 4: number analyzed (Participants) | 61 | 63
  Change at Week 4 | -0.03 (0.070) | 0.91 (0.117)
  Change at Week 12: number analyzed (Participants) | 61 | 64
  Change at Week 12 | 0.11 (0.082) | 0.70 (0.107)
  Change at Week 22: number analyzed (Participants) | 63 | 62
  Change at Week 22 | 0.02 (0.069) | 1.01 (0.123)
  Change at Week 24: number analyzed (Participants) | 62 | 66
  Change at Week 24 | 0.07 (0.071) | 0.51 (0.093)
  Change at Week 48: number analyzed (Participants) | 62 | 61
  Change at Week 48 | 0.55 (0.087) | 0.48 (0.091)
  Change at Week 60: number analyzed (Participants) | 58 | 58
  Change at Week 60 | 0.57 (0.097) | 0.43 (0.086)
  Change at Week 72: number analyzed (Participants) | 57 | 57
  Change at Week 72 | 0.55 (0.086) | 0.43 (0.091)
  Change at Week 84: number analyzed (Participants) | 57 | 56
  Change at Week 84 | 0.49 (0.078) | 0.42 (0.092)
  Change at Week 96: number analyzed (Participants) | 58 | 57
  Change at Week 96 | 0.29 (0.086) | 0.46 (0.084)

25. Secondary Outcome: Percent Change From Baseline Over Time in TmP/GFR
Description: The GEE Estimates are from the GEE model which includes the percent change from baseline for TmP/GFR as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of TmP/GFR as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 2, 4, 12, 22, 24, 48, 60, 72, 84, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 63 | 66
percentage change
  Change at Week 2: number analyzed (Participants) | 60 | 60
  Change at Week 2 | -2.15 (4.515) | 100.10 (7.222)
  Change at Week 4: number analyzed (Participants) | 61 | 63
  Change at Week 4 | -2.73 (4.416) | 56.53 (6.816)
  Change at Week 12: number analyzed (Participants) | 61 | 64
  Change at Week 12 | 6.28 (4.900) | 43.65 (6.206)
  Change at Week 22: number analyzed (Participants) | 63 | 62
  Change at Week 22 | 1.38 (4.252) | 62.38 (7.144)
  Change at Week 24: number analyzed (Participants) | 62 | 66
  Change at Week 24 | 3.63 (4.460) | 33.02 (5.464)
  Change at Week 48: number analyzed (Participants) | 62 | 61
  Change at Week 48 | 35.52 (5.390) | 31.02 (5.489)
  Change at Week 60: number analyzed (Participants) | 58 | 58
  Change at Week 60 | 37.13 (5.855) | 27.49 (5.002)
  Change at Week 72: number analyzed (Participants) | 57 | 57
  Change at Week 72 | 35.89 (5.492) | 28.98 (5.513)
  Change at Week 84: number analyzed (Participants) | 57 | 56
  Change at Week 84 | 33.15 (4.924) | 27.69 (5.527)
  Change at Week 96: number analyzed (Participants) | 58 | 57
  Change at Week 96 | 19.95 (5.417) | 29.67 (4.759)

26. Secondary Outcome: Change From Baseline Over Time in Tubular Reabsorption of Phosphate (TRP)
Description: The GEE Estimates are from the GEE model which includes the change from baseline for TRP as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of TRP as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 2, 4, 12, 22, 24, 48, 60, 72, 84, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: fraction of phosphate reabsorbed
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 64 | 67
fraction of phosphate reabsorbed
  Change at Week 2: number analyzed (Participants) | 62 | 63
  Change at Week 2 | -0.02 (0.013) | 0.07 (0.008)
  Change at Week 4: number analyzed (Participants) | 63 | 65
  Change at Week 4 | -0.03 (0.012) | 0.03 (0.009)
  Change at Week 12: number analyzed (Participants) | 62 | 64
  Change at Week 12 | -0.00 (0.010) | 0.04 (0.008)
  Change at Week 22: number analyzed (Participants) | 63 | 64
  Change at Week 22 | -0.01 (0.009) | 0.05 (0.011)
  Change at Week 24: number analyzed (Participants) | 63 | 67
  Change at Week 24 | -0.02 (0.012) | 0.03 (0.009)
  Change at Week 48: number analyzed (Participants) | 64 | 63
  Change at Week 48 | 0.02 (0.012) | 0.03 (0.009)
  Change at Week 60: number analyzed (Participants) | 60 | 60
  Change at Week 60 | 0.03 (0.009) | 0.02 (0.009)
  Change at Week 72: number analyzed (Participants) | 60 | 59
  Change at Week 72 | 0.02 (0.011) | 0.02 (0.011)
  Change at Week 84: number analyzed (Participants) | 58 | 58
  Change at Week 84 | 0.02 (0.010) | 0.01 (0.012)
  Change at Week 96: number analyzed (Participants) | 59 | 58
  Change at Week 96 | -0.01 (0.014) | 0.03 (0.009)

27. Secondary Outcome: Percent Change From Baseline Over Time in TRP
Description: The GEE Estimates are from the GEE model which includes the percent change from baseline for TRP as the dependent variable, region, visit, treatment, actual randomization stratification and visit by treatment as fixed factors, and baseline of TRP as a covariate, with compound symmetry covariance structure.
Time Frame: Baseline, Weeks 2, 4, 12, 22, 24, 48, 60, 72, 84, 96
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Burosumab 1 mg/kg
Number analyzed (Participants) | 64 | 67
percentage change
  Change at Week 2: number analyzed (Participants) | 62 | 63
  Change at Week 2 | -2.00 (1.530) | 9.81 (1.111)
  Change at Week 4: number analyzed (Participants) | 63 | 65
  Change at Week 4 | -3.75 (1.486) | 4.86 (1.114)
  Change at Week 12: number analyzed (Participants) | 62 | 64
  Change at Week 12 | 0.56 (1.261) | 5.45 (1.079)
  Change at Week 22: number analyzed (Participants) | 63 | 64
  Change at Week 22 | -0.01 (1.163) | 7.03 (1.451)
  Change at Week 24: number analyzed (Participants) | 63 | 67
  Change at Week 24 | -1.56 (1.579) | 4.21 (1.141)
  Change at Week 48: number analyzed (Participants) | 64 | 63
  Change at Week 48 | 3.95 (1.547) | 4.70 (1.183)
  Change at Week 60: number analyzed (Participants) | 60 | 60
  Change at Week 60 | 3.99 (1.096) | 3.00 (1.123)
  Change at Week 72: number analyzed (Participants) | 60 | 59
  Change at Week 72 | 3.90 (1.427) | 3.24 (1.414)
  Change at Week 84: number analyzed (Participants) | 58 | 58
  Change at Week 84 | 3.78 (1.276) | 1.97 (1.516)
  Change at Week 96: number analyzed (Participants) | 59 | 58
  Change at Week 96 | -0.09 (1.582) | 4.44 (1.116)

28. Secondary Outcome: Percentage of Participants Achieving Mean Serum Phosphorus Levels Above the LLN (2.5 mg/dL [0.81 mmol/L]) at the End of the Dosing Cycle, as Averaged Across Dose Cycles Between Baseline and Week 24
Time Frame: Baseline through Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Burosumab
Number analyzed (Participants) | 66 | 68
percentage of participants | 6.1 [2.4 to 14.6] | 67.6 [55.8 to 77.6]

29. Secondary Outcome: Change From Baseline in Serum Phosphorus at Each Mid-Point of Dosing Cycle, as Averaged Across Dose Cycles Between Baseline and Week 24
Time Frame: Baseline through Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Burosumab
Number analyzed (Participants) | 66 | 68
mg/dL | 0.16 (0.272) | 1.21 (0.513)

30. Secondary Outcome: Percent Change From Baseline in Serum Phosphorus at Each Mid-Point of Dosing Cycle, as Averaged Across Dose Cycles Between Baseline and Week 24
Time Frame: Baseline through Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Burosumab
Number analyzed (Participants) | 66 | 68
percentage change | 9.85 (15.292) | 61.44 (28.961)

31. Secondary Outcome: Change From Baseline in Serum Phosphorus at Each End of Dosing Cycle, as Averaged Across Dose Cycles Between Baseline and Week 24
Time Frame: Baseline through Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Burosumab
Number analyzed (Participants) | 66 | 68
mg/dL | 0.13 (0.265) | 0.69 (0.392)

32. Secondary Outcome: Percent Change From Baseline in Serum Phosphorus at Each End of Dosing Cycle, as Averaged Across Dose Cycles Between Baseline and Week 24
Time Frame: Baseline through Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | Burosumab
Number analyzed (Participants) | 66 | 68
percentage change | 7.83 (14.755) | 35.18 (20.731)

33. Secondary Outcome: Time-Adjusted Area Under the Curve (AUC) of Serum Phosphorus Between Baseline and Week 24
Time Frame: Baseline through Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Burosumab
Number analyzed (Participants) | 66 | 68
mg/dL | 2.08 (0.292) | 3.08 (0.477)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the end of study plus 4 weeks (+ 5 days). Mean (SE) duration of exposure to burosumab for all periods combined through EOS II was 771.3 (21.97) days (range: 167 - 957) in the burosumab->burosumab group and 625.7 (19.40) days (range: 165 - 844) in the placebo->burosumab group.
Groups:
- Placebo (DB Period): SC injection of placebo Q4W for 24 weeks (double-blind placebo-controlled Treatment Period)
- Placebo -> Burosumab (OL Period): SC injection of placebo Q4W for 24 weeks (double-blind placebo-controlled Treatment Period), SC injection of burosumab 1 mg/kg Q4W for 24 weeks (open-label Treatment Continuation Period), SC injection of burosumab 1 mg/kg Q4W for 48 weeks (open label Treatment Extension Period I), and SC injection of burosumab 1 mg/kg Q4W up to 53 weeks (open-label Treatment Extension Period II [US only]).
- Burosumab -> Burosumab (Combined DB and OL Period): SC injection of 1.0 mg/kg burosumab Q4W for 24 weeks (double-blind placebo-controlled Treatment Period), SC injection of burosumab 1 mg/kg Q4W for 24 weeks (open-label Treatment Continuation Period), SC injection of burosumab 1 mg/kg Q4W for 48 weeks (open-label Treatment Extension Period I), and SC injection of burosumab 1 mg/kg Q4W up to 53 weeks (open-label Treatment Extension Period II [US only]).
- Total Burosumab (Combined DB and OL Period): SC injection of 1.0 mg/kg burosumab at any time during the study.
Arm/Group | Placebo (DB Period) | Placebo -> Burosumab (OL Period) | Burosumab -> Burosumab (Combined DB and OL Period) | Total Burosumab (Combined DB and OL Period)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66 | 1/68 | 1/134
Serious Adverse Events (participants affected / at risk) | 1/66 | 10/66 | 12/68 | 22/134
Other Adverse Events (participants affected / at risk) | 57/66 | 63/66 | 68/68 | 131/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (DB Period) (N=66) | Placebo -> Burosumab (OL Period) (N=66) | Burosumab -> Burosumab (Combined DB and OL Period) (N=68) | Total Burosumab (Combined DB and OL Period) (N=134)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Periodontal Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Peritoneal Adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1
Medical Device Site Infection (Infections and infestations) | 0 | 0 | 1 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural Nausea (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural Vomiting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Joint Range Of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Knee Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Parathyroid Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Cerebrospinal Fluid Leakage (Nervous system disorders) | 0 | 0 | 1 | 1
Cervical Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 0 | 2 | 2
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1
Partial Seizures (Nervous system disorders) | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (DB Period) (N=66) | Placebo -> Burosumab (OL Period) (N=66) | Burosumab -> Burosumab (Combined DB and OL Period) (N=68) | Total Burosumab (Combined DB and OL Period) (N=134)
Vertigo (Ear and labyrinth disorders) | 1 | 4 | 3 | 7
Hyperparathyroidism Secondary (Endocrine disorders) | 0 | 3 | 4 | 7
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 3 | 4 | 7
Abdominal Pain (Gastrointestinal disorders) | 2 | 2 | 6 | 8
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 6 | 3 | 9
Constipation (Gastrointestinal disorders) | 0 | 4 | 10 | 14
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 13 | 18
Nausea (Gastrointestinal disorders) | 6 | 5 | 11 | 16
Toothache (Gastrointestinal disorders) | 1 | 10 | 12 | 22
Vomiting (Gastrointestinal disorders) | 2 | 4 | 6 | 10
Asthenia (General disorders) | 2 | 1 | 5 | 6
Fatigue (General disorders) | 7 | 14 | 16 | 30
Injection Site Erythema (General disorders) | 2 | 6 | 6 | 12
Injection Site Pruritus (General disorders) | 0 | 8 | 3 | 11
Injection Site Reaction (General disorders) | 2 | 8 | 7 | 15
Pain (General disorders) | 6 | 9 | 12 | 21
Pyrexia (General disorders) | 0 | 4 | 5 | 9
Seasonal Allergy (Immune system disorders) | 1 | 6 | 5 | 11
Bronchitis (Infections and infestations) | 1 | 6 | 4 | 10
Gastroenteritis (Infections and infestations) | 2 | 4 | 2 | 6
Influenza (Infections and infestations) | 3 | 6 | 9 | 15
Nasopharyngitis (Infections and infestations) | 6 | 24 | 28 | 52
Oral Herpes (Infections and infestations) | 0 | 4 | 4 | 8
Pharyngitis (Infections and infestations) | 1 | 0 | 4 | 4
Rhinitis (Infections and infestations) | 1 | 4 | 1 | 5
Sinusitis (Infections and infestations) | 2 | 2 | 6 | 8
Tooth Abscess (Infections and infestations) | 6 | 5 | 19 | 24
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 2 | 12 | 14
Urinary Tract Infection (Infections and infestations) | 4 | 6 | 5 | 11
Contusion (Injury, poisoning and procedural complications) | 1 | 5 | 4 | 9
Fall (Injury, poisoning and procedural complications) | 0 | 7 | 6 | 13
Ligament Sprain (Injury, poisoning and procedural complications) | 6 | 2 | 4 | 6
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 6 | 9 | 15
Blood 25-Hydroxycholecalciferol Decreased (Investigations) | 1 | 3 | 6 | 9
Blood Glucose Increased (Investigations) | 0 | 1 | 5 | 6
Blood Parathyroid Hormone Increased (Investigations) | 1 | 1 | 5 | 6
Blood Pressure Increased (Investigations) | 1 | 1 | 6 | 7
Lipase Increased (Investigations) | 0 | 0 | 4 | 4
Vitamin D Decreased (Investigations) | 0 | 9 | 8 | 17
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 4 | 4
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 5
Vitamin D Deficiency (Metabolism and nutrition disorders) | 3 | 7 | 15 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 23 | 27 | 50
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 17 | 18 | 35
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 8 | 14
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4 | 8
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 7 | 5 | 12
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 9 | 11 | 20
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 6 | 8
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 3 | 7
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 | 10 | 12 | 22
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 3 | 4 | 4 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 8 | 13
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 3 | 8
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 10 | 10 | 18 | 28
Dizziness (Nervous system disorders) | 4 | 5 | 11 | 16
Headache (Nervous system disorders) | 5 | 18 | 22 | 40
Hypoaesthesia (Nervous system disorders) | 1 | 3 | 7 | 10
Migraine (Nervous system disorders) | 1 | 2 | 7 | 9
Restless Legs Syndrome (Nervous system disorders) | 5 | 10 | 11 | 21
Depression (Psychiatric disorders) | 1 | 3 | 9 | 12
Insomnia (Psychiatric disorders) | 1 | 6 | 9 | 15
Nephrocalcinosis (Renal and urinary disorders) | 0 | 4 | 2 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 11 | 10 | 21
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 5 | 10
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 4 | 12
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 6
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 4 | 5
Hot Flush (Vascular disorders) | 0 | 2 | 6 | 8
Hypertension (Vascular disorders) | 2 | 5 | 8 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.